CLINICAL TRIAL: NCT02410590
Title: Randomized, Parallel Group, Controlled Trial to Compare Two Different "NMB + Reversal" Strategies in Adult Obese Patients Undergoing Laparoscopic Abdominal Surgery
Brief Title: Rocuronium + Sugammadex vs. Succinylcholine + Cisatracurium + Neostigmine/Atropine in Obese Participants (MK-8616-104)
Acronym: BENN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 8616-104; 2013-004423-36 (EudraCT Number)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium; Sugammadex; cisatracurium; Neostigmine; Atropine; Succinylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rocuronium + Sugammadex (Experimental): Participants will receive rocuronium administered at a dosage adequate to make intubation possible and provide deep NMB (defined as no response to train-of-four stimulation but at least one response to five post-tetanic count [PTC]) for the duration of surgery, until the end of the procedure. Sugammadex will be administered to participants once at a dosage of 4 mg/kg real body weight (RBW) IV at the end of surgical procedure. Sugammadex will be used as the only reversal drug in all participants who receive rocuronium as a neuromuscular blocker.
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- Succinylcholine + Cisatracurium + Neostigmine/Atropine (Active Comparator): After receiving succinylcholine 1.0 mg/kg RBW for intubation, participants will receive cisatracurium administered at dosage adequate to have a moderate NMB (defined as a target of TOF ratio = 10% with a range: 2-3 twitches to TOF ratio of 20%) for the duration of surgery, until the end of the procedure. Neostigmine/Atropine will be administered to participants once at respective dosage of 0.05 mg/kg RBW and 0.01 mg/kg RBW at least after the reappearance of T2 after surgery completion. The maximum allowed dosage for Neostigmine is 5 mg. Neostigmine will be used as only reversal drug in all participants who received Cisatracurium as neuromuscular blocker.
  Interventions: Drug: Cisatracurium; Drug: Neostigmine/Atropine; Drug: Succinylcholine

INTERVENTIONS:
Drug: Rocuronium
  Arms: Rocuronium + Sugammadex
Drug: Sugammadex
  Arms: Rocuronium + Sugammadex
Drug: Cisatracurium
  Arms: Succinylcholine + Cisatracurium + Neostigmine/Atropine
Drug: Neostigmine/Atropine
  Arms: Succinylcholine + Cisatracurium + Neostigmine/Atropine
Drug: Succinylcholine
  Arms: Succinylcholine + Cisatracurium + Neostigmine/Atropine

SUMMARY:
The primary objective of this trial is to compare the preference between two strategies of neuromuscular blocking (NMB) / reversal in adult obese patients undergoing laparoscopic abdominal surgery: Rocuronium + Sugammadex versus Succinylcholine + Cisatracurium + Neostigmine/Atropine. This will be done evaluating the average verbal numerical scale (VNS) scores obtained from surgeons blinded to the drugs administered. The primary hypothesis is that the strategy "Rocuronium + Sugammadex" provides a better surgical visual field in obese participants undergoing laparoscopic abdominal surgery than the strategy "Succinylcholine + Cisatracurium + Neostigmine/Atropine" as measured by VNS scores.

ELIGIBILITY:
Inclusion Criteria:

* must be obese, with a Body Mass Index ≥30.0 to ≤50.
* must be scheduled to undergo an elective abdominal laparoscopic surgery, under general anesthesia. (Participants are expected to remain in the hospital for at least 24 hours following surgical procedure.)
* must be categorized as American Society of Anesthesiologists (ASA) Class 1, 2, or 3.
* clinical laboratory tests within normal limits or clinically acceptable to the investigator/sponsor.
* sexually active females of child-bearing potential must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for the 30 days after stopping the medication. Medically accepted methods of contraception include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, inert or copper-containing IUD, hormone-releasing IUD, systemic hormonal contraceptive, and surgical sterilization (eg, hysterectomy or tubal ligation). Postmenopausal women are not required to use contraception. Postmenopausal is defined as at least 12 consecutive months without a spontaneous menstrual period. Each sexually active male subject with a female partner(s) of childbearing potential must also provide written informed consent to provide information regarding any pregnancy.

Exclusion Criteria:

* has anatomical malformations that may lead to difficult intubation.
* is known or suspected to have neuromuscular disorders that may affect NMB and/or trial assessments.
* history of previous abdominal laparoscopy procedures.
* must not currently (within past 6 months) meet DSM-IV-TR criteria for substance abuse or dependence (excluding nicotine).
* history of a chronic pain condition (requiring continuous/daily pain medication prior to surgery).
* females who have given birth to one or more children in the last 12 months, or are pregnant or intend to become pregnant between randomization and >Day 30 pregnancy follow-up contact [premenopausal female of childbearing potential].
* evidence of acute cholecystitis.
* dialysis-dependency or suspected of having severe renal insufficiency (defined as estimated creatinine clearance of <30 mL/min).
* significant hepatic dysfunction that would prevent participation in the trial, based on the summary of product characteristics of the study drugs.
* history of or family history of malignant hyperthermia.
* known allergy to trial treatments (rocuronium, sugammadex, succinylcholine, cisatracurium, neostigmine, atropine) or their excipients, to opioids/opiates, or other medication used during general anesthesia.
* expected transfer to intensive care unit after surgery.
* must continue to receive toremifene or fusidic acid during the trial.
* has participated in another clinical trial within 30 days of signing the informed consent form of the current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Number of Surgeons who prefer Rocuronium + Sugammadex vs. Succinylcholine + Cisatracurium + Neostigmine/Atropine for neuromuscular blocking/reversal in obese participants undergoing laparoscopic abdominal surgery | Up to 1 hour after end of surgery

SECONDARY OUTCOMES:
Time elapsed from end of surgery to extubation | Up to 1 hour after end of surgery
Time elapsed from start of reversal drug administration to train-of-four (TOF) ratio ≥0.9 | Up to 1 hour after start of reversal drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC